CLINICAL TRIAL: NCT02847897
Title: Evaluation of the Safety and Efficacy of Carbon Dioxide (CO2) Acupulse Laser for the Treatment of Vaginal Prolapse in Women.
Brief Title: Evaluation of Safety and Efficacy of Carbon Dioxide (CO2) Acupulse Laser Treatment on Vaginal Elasticity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Dr. Roy Lauterbach, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0217-16-RMB
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Exposure Laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CO2 AcuPulse Laser treatment (Experimental): Subjects with vulvovaginal atrophy intended to receive 3 treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.
  Interventions: Device: CO2 AcuPulse Laser

INTERVENTIONS:
Device: CO2 AcuPulse Laser — Each subject will receive 3 treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.

SUMMARY:
The study is intended to assess the safety and efficacy of CO2 AcuPulse laser treatment in patients with vaginal prolapse. Eligible subjects will receive 3 treatment sessions, 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.

DETAILED DESCRIPTION:
Following a screening visit, eligible subjects will be enrolled into the study. Each subject will receive 3 treatments 4 weeks apart and 3 Follow Up visits, at 1, 3, and 6 months following the last treatment.

Further demographic information and patient history will be obtained from the subjects' electronical files.

ELIGIBILITY:
Inclusion Criteria:

• Healthy post-menopausal women as defined by one of the following: A. ≥ 40 years old, last spontaneous menstrual bleeding occurred at least ≥ 12 months prior to screening B. ≥ 45 years old, does not remember the date of last spontaneous menstrual bleeding and provides lab results showing that the follicle-stimulating hormone (FSH) level is > 40 IU/L C. Underwent a hysterectomy without oophorectomy and provides lab results showing that serum FSH levels > 40IU/L D. Underwent bilateral oophorectomy at least 12 weeks prior to screening

* Presence of one or more of the prolapse related symptoms (e.g. dryness, itching, burning, dysuria or dyspareunia)
* At least 10 subjects of the sample will have symptoms of urinary stress incontinence (Stamey classification Grade =1)
* Negative urine analysis
* Normal Papanicolaou (PAP) test from the recent year
* Sexually active (having sex at least once a month) or wishing to maintain an active sexual life
* Able and willing to comply with the treatment/follow-up schedule and requirements

Exclusion Criteria:

* Vaginal Health Index Score (VHIS) < 5
* Active genital infection
* Subject presenting abnormal PAP result from the last three years with any of the following findings according to the Bethesda System (2001) classification:

A. Atypical Squamous Cells of Undetermined Significance (ASCUS with positive human papilloma virus (HPV) High Risk Positive B. Atypical Squamous Cells-cannot exclude high grade squamous intraepithelial lesion C. Atypical Glandular Cells (Endocervical, Endometrial not otherwise specified) D. Low Grade squamous intraepithelial lesion (LSIL) E. High Grade squamous intraepithelial lesion (HSIL) F. Carcinoma

* Systemic steroids use within the last 3 months
* Systemic hormonal replacement therapies within the last 3 months
* Local hormonal replacement therapies within last month
* Vaginal lubricants within 7 days prior to enrollment
* Recurring urinary tract infection or recurring infection of genital herpes or candida (> 2 episodes in the recent year)
* Pelvic organ prolapse (POP) >II according to the pelvic organ prolapse quantification system
* Transvaginal mesh implant
* Serious systemic disease or any chronic condition that could interfere with study compliance
* Taken part in a clinical trial within 30 days prior to screening.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
The change in vaginal prolapse symptoms as measured by VHI score at 3 months follow-up visit compared to baseline. | 8 months.

SECONDARY OUTCOMES:
• Prolapse symptoms improvement as evaluated by the investigator using VHI score at 1 and 6 months follow up visits compared to baseline | 8 months.
• Prolapse symptoms improvement as evaluated by the subject using Visual Analogue Scale (VAS) at 1, 3 and 6 months follow up visits compared to baseline | 8 months.
• Improvement in sexual function as evaluated by the subject Female Sexual Function Index (FSFI) at 1, 3 and 6 months follow up visits compared to baseline | 8 months.
• Improvement in urinary incontinence as evaluated by subject Incontinence Quality of Life Questionnaire (I-QOL) at 1, 3 and 6 months follow up visits compared to baseline. | 8 months.
• Improvement in prolapse grade at 1, 3 and 6 months follow up visits compared to baseline | 8 months.
• Subject satisfaction with the treatment sing a 5-point Likert scale at baseline and at 1, 3 and 6 months follow up visits | 8 months.
• Subject self- assessment of downtime related to procedure - the period of time following the procedure during which the subject felt uncomfortable/unwilling or unable to have sexual intercourse | 8 months.
• Subject assessment of pain and discomfort that is procedure related using a visual a Pain Visual Analogue Scale (VAS), evaluated at each treatment. | 8 months.
Adverse events (AE's) and serious adverse events (SAE's) | 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No